CLINICAL TRIAL: NCT04812288
Title: Oxygenation and Muscle Function's Relationship During Short Light-Intensity Exercise in Older Adults
Brief Title: Oxygenation and Muscle Function's Relationship During SLIE in Older Adults
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Fei Zhao, Student, State University of New York at Buffalo
Other Study IDs: STUDY00003426
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Oxygenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to determine the correlations between oxygenation of calf muscles and physical performance including balance, gait speed, and endurance in older adults by utilizing the NIRS device.

DETAILED DESCRIPTION:
The aim of this study is to determine the relationship between oxygenation of calf muscles and physical performance including balance, gait speed, and endurance in older adults by utilizing the NIRS device. The investigators want to determine the relationship between different types of tests and oxygenation for older adults with 4 levels of physical activity. This study will help towards identifying possible short and effective exercises for older adults with different activity levels.

ELIGIBILITY:
Inclusion Criteria:

* individuals who are 60 years old or older
* who are ambulatory with or without a mobility device
* can follow instructions without assistance

Exclusion Criteria:

* having an amputated limb
* current or uncontrolled vestibular disorders
* sensation impairment at the lower extremity
* macular degeneration disease such as glaucoma
* Parkinson's disease
* blood circulation disorders such as chronic venous insufficiency
* individuals without English proficiency

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults aged 60 and over were included.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-06-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
time to reach the minimum muscular oxygenation level (Only measure one time at a single time point, does not measure changes) | Day1
  time to reach the minimum muscular oxygenation level during bilateral heel raise test in seconds
recovery of muscular oxygenation (Only measure one time at a single time point, does not measure changes) | Day1
  the muscular oxygenation difference in percentage between the first second and the last second after finishing the bilateral heel raise test for 1 minute

SECONDARY OUTCOMES:
time to finish the Timed Up and Go test (Only measure one time at a single time point, does not measure changes) | Day1
  This test measures time in seconds to finish the Timed Up and Go test from standing from a chair, walking for 3-meter distance, turning around, going back and sitting down. Less seconds means higher mobility. Higher than 12 seconds indicates risk of falls.
Short Physical Performance Battery score (Only measure one time at a single time point, does not measure changes) | Day1
  Three parts including balance, gait speed, and chair stand test are measured. Full points of each part is 4. The score range is from 0 to 12 points. Higher score means higher physical function.
distance finished in the 2-Minute Walking test (Only measure one time at a single time point, does not measure changes) | Day1
  This test measures the maximum distance in meters covered in 2 minutes. Longer distance means better endurance.
the number of heel raise finished within one minute (Only measure one time at a single time point, does not measure changes) | Day1
  This test measures the number of heel raise that participants can complete within one minute. More heel raise times means more endurance at the calf muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Zhao, MPT, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No